CLINICAL TRIAL: NCT03524469
Title: Studying Infant Nutrition and Glycemia (SING)
Brief Title: Studying Infant Nutrition and Blood Sugar
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Bridget Young, Research Assistant Professor, University of Rochester
Other Study IDs: RSRB71535; K01DK115710 (NIH)
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — maternal blood, stool and breast milk infant urine, stool and dried blood spot card
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal weight: "Normal Weight" will be defined as pre-pregnant BMI between 18.5-23.9 kg/m2 and passing the 28 week oral glucose tolerance test.
- Insulin resistant: "Insulin Resistance" will be defined as meeting any of the following:
  * pre-pregnant BMI ≥ 28 and failed the 28 week oral glucose screening test
  * pre-pregnant BMI ≥ 28 and diagnosis of either A1 ("diet controlled") or A2 ("insulin-requiring") gestational diabetes during pregnancy, but insulin therapy discontinued after birth.
  * pre-pregnant BMI ≥ 28 and diagnosed with type 2 diabetes during pregnancy
  * pre-pregnant BMI ≥ 30, and unmediated.

SUMMARY:
The purpose of this study is to learn about how breast milk from mothers with insulin-resistance may be different. Investigators are specifically studying insulin concentrations in breast milk. Investigators are also studying how insulin in breast milk might affect a baby's intestines and pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Mothers ≥ 19 years of age
* Mothers intending to Exclusively Breastfeed for at least 5months
* Mothers comfortable with feeding their infants expressed breast milk from a bottle at 2-weeks postpartum
* Trial of labor (no scheduled C-sections)
* Singleton birth
* Healthy Infants
* "Normal Weight" will be defined as pre-pregnant BMI between 18.5-23.9 kg/m2 and passing the 28 week oral glucose tolerance test.
* "Insulin Resistance" will be defined as meeting any of the following:

  * pre-pregnant BMI ≥ 28 and failed the 28 week oral glucose screening test
  * pre-pregnant BMI ≥ 28 and diagnosis of either A1 ("diet controlled") or A2 ("insulin-requiring") gestational diabetes during pregnancy, but insulin therapy discontinued after birth.
  * pre-pregnant BMI ≥ 28 and diagnosed with type 2 diabetes during pregnancy
  * pre-pregnant BMI ≥ 30, and unmediated.

Exclusion Criteria:

* Scheduled C-sections or emergency C-sections with no labor (natural or induced)
* Maternal insulin therapy after birth
* Significant maternal health concern including type 1 diabetes, renal, kidney, thyroid, or cardiovascular disease, pre-eclampsia, or other disease.
* Delivery before 37 weeks
* Infant birth weight <2500g
* Infant medical or genetic indications that would impact normal feeding behavior, insulin signaling or growth patterns
* Infant supplementation with infant formula (glucose gel or donor milk is acceptable)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria were selected to include only healthy infants of uncomplicated pregnancy (with the exception of gestational diabetes) and normal birth weight. The criteria for insulin resistance were strategically defined to capture the insulin-resistant population which represents a large proportion of the population that are at risk for diabetes but have not yet developed the disease. Insulin therapy is an exclusion criteria because it passes through the breast milk and we are unable to distinguish endogenous maternal insulin from exogenous therapeutic insulin in breast milk samples. These criteria will minimize the risks and increase the safety of subjects.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
mean infant postprandial C peptide to creatinine ratio | 2 weeks
  Postprandial urine (60-90 minute) will be tested for C peptide and creatinine and the ratio will be calculated.

SECONDARY OUTCOMES:
mean infant insulinogenic index | 5 months
  The insulinogenic index will be measures in infant blood at 0 and 30 minutes post glucose administration. The index is the change in insulin over the change in glucose.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center of the University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No